CLINICAL TRIAL: NCT03821194
Title: The Effect of Chronic Pain Relief Over Knee Joint Area by Gua Sha Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-08-030A
Record Dates: First submitted 2018-12-20; First posted 2019-01-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pain, Chronic
Keywords: pain relief; complementary and alternative therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: chronic knee joint pain patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gua sha group (Experimental): do gua sha for the subjects
  Interventions: Other: Gua sha
- control group (Active Comparator): give hot pack for the subjects
  Interventions: Other: hot pack

INTERVENTIONS:
Other: Gua sha — Scrape the skin around the knee joint
  Arms: Gua sha group
Other: hot pack — hot pack
  Arms: control group

SUMMARY:
Objective:

A randomized, single-blind, controlled clinical trial is conducted to evaluate the effect of gua sha on the relief of chronic knee joint area pain, and to investigate the association between local skin surface and core temperature changes with chronic pain relief over knee after gua sha. Also, we want to observe the changes before and after gua sha in the local tissues of the knee joint area. We expect to provide more insights into the relevant mechanism of gua sha and relieving pain in chronic knee joint area and establish a complementary therapy for chronic knee joint pain.

Materials and Methods:

In this study, a total of 40 chronic knee joint pain participants will be recruited in the eligible conditions. After agreeing into the clinical study and signing the informed consent form, they will be randomized assigned into the treatment group (20 persons) and control group (20 people). Both groups will be tested for total of 12 days. For treatment group, 2 times of gua sha method will be applied within 12-day test period, the treatments will be on the first day and the fourth day respectively. The control group will be applied 2 times of hot pack method at same period intervals during the 12 days. Both groups will be measured the surface and core temperature of the applied site before and after each method. The visual analog scale (VAS) and the lower extremity functional scale (LEFS) and SF-12 quality of life questionnaire will be performed before and after the test. Ultrasound scans of knee will be performed before and after the test. After the data collection is completed, the analysis is performed in SPSS version 24. Student's t-test and one-way ANOVA methods will be used, with P<0.05 as a significant result.

Expected results:

To establish the positive effect of gua sha therapy to relieve the chronic knee joint pain, and use data and images to infer the mechanism of gua sha therapy on relieving chronic knee joint pain.

ELIGIBILITY:
Inclusion Criteria:

1. Those aged 20-60 years old
2. There are at least three pains in the unilateral or bilateral knee joints (up and down steps, squats, running, squatting, jumping, walking, and sedentary for a long time), and the pain lasts for at least one month.
3. Visual pain score (VAS) ≧30 (mm) for unilateral or bilateral knee joints
4. Non-steroidal anti-inflammatory drugs, analgesics, and Chinese herbal medicines for the treatment of knee joint pain
5. Non-severe degenerative arthritis (Kellgren-Lawrence scale knee arthritis grade 2 or less)

Exclusion Criteria:

1. thighs, knee joints, calf areas, those who have undergone surgery or are expected to have surgery, those who have been traumatized within the last month, and those who have wounds, ulcers, infections or other skin diseases within two weeks
2. Pregnancy
3. BMI value is greater than 27 KG/m2
4. People with cardiovascular disease or hemophilia
5. Patients with gout, rheumatism and rheumatoid arthritis
6. Diabetic patients with knee arthritis, patients with dry arthritis
7. Patients with malignant tumors
8. Those who are allergic to Vaseline products

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-09-22 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 10 Days
  To assess the pain degree. Scale: 0~100 mm, higher scores, higher pain . Counted by each time recording.
Lower Extremity Functional Scale | 10 Days
  Evaluate the functional impairment of a patient with a disorder of one or both lower extremities.
  Scale: 0~80, higher scores, higher lower extremity function Counted by each time recording.
Short Form-12 Health Survey | 3 Days
  Evaluate the health-related quality of life, use SF-12 questionnaire. Scale: 0~100, higher scores, better life quality. Counted by each time recording and using mode conversion to get final scale.

SECONDARY OUTCOMES:
Ultrasound scans of knee | 3 Days
  To observe the tissue of knee joint, compare quadriceps muscle changes and tendon thickness before and after treatment.
  No special measure, just take picture of ultrasound scans and compare the picture.
surface temperature | 2 hours
  To evaluate the knee joint surface temperature before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Pey Chen, MD, Study Chair — Center for Traditional Medicine, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel DR, Villalobos A. Evaluation and management of knee pain in young athletes: overuse injuries of the knee. Transl Pediatr. 2017 Jul;6(3):190-198. doi: 10.21037/tp.2017.04.05. PMID 28795010
- [Background] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Background] Werner S. Anterior knee pain: an update of physical therapy. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2286-94. doi: 10.1007/s00167-014-3150-y. Epub 2014 Jul 6. PMID 24997734
- [Background] Iagnocco A, Naredo E. Osteoarthritis: research update and clinical applications. Rheumatology (Oxford). 2012 Dec;51 Suppl 7:vii2-5. doi: 10.1093/rheumatology/kes328. PMID 23230089
- [Background] Cowan DT, Fitzpatrick JM, Roberts JD, While AE, Baldwin J. The assessment and management of pain among older people in care homes: current status and future directions. Int J Nurs Stud. 2003 Mar;40(3):291-8. doi: 10.1016/s0020-7489(02)00087-1. PMID 12605951
- [Background] MacPherson H, Maschino AC, Lewith G, Foster NE, Witt CM, Vickers AJ; Acupuncture Trialists' Collaboration. Characteristics of acupuncture treatment associated with outcome: an individual patient meta-analysis of 17,922 patients with chronic pain in randomised controlled trials. PLoS One. 2013 Oct 11;8(10):e77438. doi: 10.1371/journal.pone.0077438. eCollection 2013. PMID 24146995
- [Background] WHO. WHO Traditional Medicine Strategy 2014-2023. WHO Library Cataloguing-inPublication Data. 2013.
- [Background] Sun C, Desai GJ, Pucci DS, Jew S. Musculoskeletal disorders: does the osteopathic medical profession demonstrate its unique and distinctive characteristics? J Am Osteopath Assoc. 2004 Apr;104(4):149-55. PMID 15127982
- [Background] Nielsen A, Knoblauch NT, Dobos GJ, Michalsen A, Kaptchuk TJ. The effect of Gua Sha treatment on the microcirculation of surface tissue: a pilot study in healthy subjects. Explore (NY). 2007 Sep-Oct;3(5):456-66. doi: 10.1016/j.explore.2007.06.001. PMID 17905355
- [Background] Nielsen A. Gua sha research and the language of integrative medicine. J Bodyw Mov Ther. 2009 Jan;13(1):63-72. doi: 10.1016/j.jbmt.2008.04.045. Epub 2008 Jul 17. PMID 19118794
- [Background] Hautman MA. Self-care responses to respiratory illnesses among Vietnamese. West J Nurs Res. 1987 May;9(2):223-43. doi: 10.1177/019394598700900205. No abstract available. PMID 3649128
- [Background] Braun M, Schwickert M, Nielsen A, Brunnhuber S, Dobos G, Musial F, Ludtke R, Michalsen A. Effectiveness of traditional Chinese "gua sha" therapy in patients with chronic neck pain: a randomized controlled trial. Pain Med. 2011 Mar;12(3):362-9. doi: 10.1111/j.1526-4637.2011.01053.x. Epub 2011 Jan 28. PMID 21276190
- [Background] Yuen JWM, Tsang WWN, Tse SHM, Loo WTY, Chan ST, Wong DLY, Chung HHY, Tam JKK, Choi TKS, Chiang VCL. The effects of Gua sha on symptoms and inflammatory biomarkers associated with chronic low back pain: A randomized active-controlled crossover pilot study in elderly. Complement Ther Med. 2017 Jun;32:25-32. doi: 10.1016/j.ctim.2017.03.010. Epub 2017 Mar 21. PMID 28619301
- [Background] Lauche R, Wubbeling K, Ludtke R, Cramer H, Choi KE, Rampp T, Michalsen A, Langhorst J, Dobos GJ. Randomized controlled pilot study: pain intensity and pressure pain thresholds in patients with neck and low back pain before and after traditional East Asian "gua sha" therapy. Am J Chin Med. 2012;40(5):905-17. doi: 10.1142/S0192415X1250067X. PMID 22928824
- [Background] Wang Y, Yang L, Yang J, Yang J, Liu Z, Chen F, Liu D, Yuan H, Wang L. Curative effect of scraping therapies on lumbar muscle strain. J Tradit Chin Med. 2013 Aug;33(4):455-60. doi: 10.1016/s0254-6272(13)60148-x. PMID 24187865
- [Background] Chiu JY, Gau ML, Kuo SY, Chang YH, Kuo SC, Tu HC. Effects of Gua-Sha therapy on breast engorgement: a randomized controlled trial. J Nurs Res. 2010 Mar;18(1):1-10. doi: 10.1097/JNR.0b013e3181ce4f8e. PMID 20220605
- [Background] Chan ST, Yuen JW, Gohel MD, Chung CP, Wong HC, Kwong KK. Guasha-induced hepatoprotection in chronic active hepatitis B: a case study. Clin Chim Acta. 2011 Aug 17;412(17-18):1686-8. doi: 10.1016/j.cca.2011.05.009. Epub 2011 May 13. PMID 21616064
- [Background] Tu WZ, Cheng RD, Hu J, Wang JZ, Lin HY, Zou EM, Wang WS, Lou XF, Jiang SH. Combination treatment with Gua Sha and Blood-letting causes attenuation of systemic inflammation, activated coagulation, tissue ischemia and injury during heatstroke in rats. Chin J Integr Med. 2015 Aug;21(8):610-7. doi: 10.1007/s11655-014-1816-4. Epub 2014 Aug 7. PMID 25098257
- [Background] Kwong KK, Kloetzer L, Wong KK, Ren JQ, Kuo B, Jiang Y, Chen YI, Chan ST, Young GS, Wong ST. Bioluminescence imaging of heme oxygenase-1 upregulation in the Gua Sha procedure. J Vis Exp. 2009 Aug 28;(30):1385. doi: 10.3791/1385. PMID 19718012
- [Background] Xu QY, Yang JS, Yang L, Wang YY. Effects of different scraping techniques on body surface blood perfusion volume and local skin temperature of healthy subjects. J Tradit Chin Med. 2011 Dec;31(4):316-20. doi: 10.1016/s0254-6272(12)60011-9. PMID 22462238
- [Background] Jones BQ, Covey CJ, Sineath MH Jr. Nonsurgical Management of Knee Pain in Adults. Am Fam Physician. 2015 Nov 15;92(10):875-83. PMID 26554281
- [Background] Simon LS. Nonsteroidal anti-inflammatory drugs and their risk: a story still in development. Arthritis Res Ther. 2013;15 Suppl 3(Suppl 3):S1. doi: 10.1186/ar4173. Epub 2013 Jul 24. PMID 24267149
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543